CLINICAL TRIAL: NCT06068452
Title: Clinical Effectiveness of Pre-operative Cardiopulmonary Exercise Testing (CPET) in Predicting Post-operative Morbidity and Mortality After Pancreatoduodenectomy- A Retrospective Cohort Study
Brief Title: Role of Pre-operative CPET in Pancreatoduodenectomy
Acronym: WHIPPLES
Status: Completed | Type: Observational
Sponsor: East Lancashire Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Meghana Taggarsi, Principal Investigator, East Lancashire Hospitals NHS Trust
Other Study IDs: 2021/010; 284588 (Other: Health Research Authority)
Record Dates: First submitted 2023-09-21; First posted 2023-10-05 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Cancer; Periampullary Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A clinical database has been prospectively maintained by the investigators, with details of pancreatic resections since January 2016. It includes pre-operative details, details of multidisciplinary team (MDT) meeting, details of pre-operative biliary stenting, intra-operative details, post-operative morbidity and mortality, details of histopathological diagnosis, recurrence and survival. Data was collected onto the database (excel sheet) from trust data software, clinic letters, Somerset Cancer registry and clinical portal.

DETAILED DESCRIPTION:
Retrospective analysis of prospectively maintained database. A clinical database has been prospectively maintained by the investigators, with details of pancreatic resections since January 2016. It includes pre-operative details, details of multidisciplinary team (MDT) meeting, details of pre-operative biliary stenting, intra-operative details, post-operative morbidity and mortality, details of histopathological diagnosis, recurrence and survival. Data was collected onto the database (excel sheet) from trust data software, clinic letters, Somerset Cancer registry and clinical portal.

Specific CPET data to be collected:

1. Exercise induced ST ischaemia- yes/no
2. VO2 peak: actual and predicted
3. Anaerobic threshold
4. VE/VCO2
5. Pulmonary function test- normal/ obstructive/ restrictive
6. Duration of pedalling bike
7. 30 day predicted risk
8. Completed the test - yes/no
9. Reason for incomplete test The CPET specific data will be collated from clinic letters, MDT meeting outcomes and CPET reports stored in hospital drive (access limited to anaesthetists only presently).

Data analysis will be done using IBM SPSS version 25. Investigators plan to use parametric and non-parametric tests and binary logistic regression analyses to compare predicted to actual mortality and morbidity, between the patients who have had CPET and those who have not.

6 STUDY SETTING: This is a single centre study, to be done at, Royal Blackburn Hospital, East Lancashire Hospitals NHS trust, a District general Hospital in North of England. The study will be carried out in the department of General and HPB surgery, in liaise with Department of anaesthesia. This is the HPB referral centre for Lancashire and South Cumbria and incorporates patients referred for pancreatic surgery from three hospital trusts (Lancashire Teaching, University Hospital Morecambe Bay and Blackpool Teaching Hospitals). The data will be stored in the trust computer system, using a password protected excel sheet. The investigators responsible for the study only, will be provided with access to the database.

ELIGIBILITY:
Inclusion Criteria:

* All pancreatic resections during the study period, performed for:

  * Cholangiocarcinoma
  * Duodenal and periampullary tumors
  * Pancreatic tumors
* All the patients in the database who have undergone Whipple (pancreatoduodenectomy)

Exclusion Criteria:

* Duodenal or gastric resections, not in conjunction with pancreatic resections
* Distal pancreatectomy
* Partial excision
* Enucleation of lesions
* Open and close when inoperable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be identified by database search from April 2016 to March 2020, online records, clinical portal, Somerset cancer registry. Duplicates will be removed, cases will be screened. All the patients who have undergone pancreatic resections for preoperative diagnosis of cholangiocarcinoma, duodenal and periampullary tumors and pancreatic tumors, which includes pancreatoduodenectomy, during the study period, irrespective of age and comorbidities will be included in the study. The patients who have undergone pancreatic resections other than pancreatoduodenectomy will be excluded. P-Possum and CPET specific data will be collected retrospectively, for predicted morbidity and mortality.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Testing (CPET)/ Portsmouth - Physiological and Operative Severity Score for the enumeration of Mortality and morbidity (P-POSSUM) predicted mortality versus actual 30 day mortality | 30 days
  Primary outcome is to compare predicted mortality by cardiopulmonary Exercise Testing (CPET)/ Portsmouth - Physiological and Operative Severity Score for the enumeration of Mortality and morbidity (P-Possum) score versus actual 30 day mortality, post-operatively.
  P-POSSUM is a scoring system for general elective and emergency surgeries which takes into account various physiological and operative parameters to calculate risk of morbidity and mortality in terms of percentages. The risk can range between 0 to 100%. The higher the percentage worse is the predicted outcome.

SECONDARY OUTCOMES:
Cardiopulmonary Exercise Testing (CPET) / Portsmouth - Physiological and Operative Severity Score for the enumeration of Mortality and morbidity (P-POSSUM) predicted morbidity versus actual post-operative morbidity | 90 days
  Secondary outcome is to compare predicted morbidity by cardiopulmonary Exercise Testing (CPET) /Portsmouth - Physiological and Operative Severity Score for the enumeration of Mortality and morbidity (P-Possum) score versus actual morbidity, post-operatively.
  P-POSSUM is a scoring system for general elective and emergency surgeries which takes into account various physiological and operative parameters to calculate risk of morbidity and mortality in terms of percentages. The risk can range between 0 to 100%. The higher the percentage worse is the predicted outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Ms Sultana, Principal Investigator — East Lancashire NHS Hospitals Trust; Meghana Ms Taggarsi, Principal Investigator — East Lancashire NHS Hospitals Trust
Locations (1):
- East Lancashire Hospitals NHS Trust, Blackburn, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Consent not obtained from participants for use of their data in future research

REFERENCES:
- [Result] Wu JM, Kuo TC, Chen HA, Wu CH, Lai SR, Yang CY, Hsu SY, Ho TW, Liao WC, Tien YW. Randomized trial of oral versus enteral feeding for patients with postoperative pancreatic fistula after pancreatoduodenectomy. Br J Surg. 2019 Feb;106(3):190-198. doi: 10.1002/bjs.11087. PMID 30724356
- [Result] Levett DZH, Jack S, Swart M, Carlisle J, Wilson J, Snowden C, Riley M, Danjoux G, Ward SA, Older P, Grocott MPW; Perioperative Exercise Testing and Training Society (POETTS). Perioperative cardiopulmonary exercise testing (CPET): consensus clinical guidelines on indications, organization, conduct, and physiological interpretation. Br J Anaesth. 2018 Mar;120(3):484-500. doi: 10.1016/j.bja.2017.10.020. Epub 2017 Nov 24. PMID 29452805
- [Result] Chandrabalan VV, McMillan DC, Carter R, Kinsella J, McKay CJ, Carter CR, Dickson EJ. Pre-operative cardiopulmonary exercise testing predicts adverse post-operative events and non-progression to adjuvant therapy after major pancreatic surgery. HPB (Oxford). 2013 Nov;15(11):899-907. doi: 10.1111/hpb.12060. Epub 2013 Feb 20. PMID 23458160
- [Result] Junejo MA, Mason JM, Sheen AJ, Bryan A, Moore J, Foster P, Atkinson D, Parker MJ, Siriwardena AK. Cardiopulmonary exercise testing for preoperative risk assessment before pancreaticoduodenectomy for cancer. Ann Surg Oncol. 2014 Jun;21(6):1929-36. doi: 10.1245/s10434-014-3493-0. Epub 2014 Jan 30. PMID 24477709

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT06068452/Prot_SAP_000.pdf